CLINICAL TRIAL: NCT04104594
Title: Olfaction and Inflammation in Chronic Rhinosinusitis With Nasal Polyps
Acronym: OIPN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The laboratory in which the analyses on nasosinusal polyposis were to be carried out did not want to continue the research on this subject, so it was decided to stop this study prematurely.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19CH099; 2019-A01625-52 (Other: ANSM)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Nasal Polyps; Chronic Rhinosinusitis With Nasal Polyps; Olfaction Disorders
Keywords: TNF alpha
MeSH Terms: conditions — Nasal Polyps; Olfaction Disorders | interventions — Smell; Sino-Nasal Outcome Test

STUDY DESIGN:
Intervention Model Description: control and patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with chronic rhinosinusitis with nasal polyps (Experimental)
  Interventions: Diagnostic Test: Sniffin Stick Test; Other: numerical evaluation scale for olfaction; Other: numerical evaluation scale for nasal obstruction; Other: nasal outcome test; Biological: dosage of 17 cytokines
- Patients with an indication for septoplasty = control group (Other)
  Interventions: Diagnostic Test: Sniffin Stick Test; Other: nasal outcome test; Biological: dosage of 17 cytokines

INTERVENTIONS:
Diagnostic Test: Sniffin Stick Test — The test consists of odorous rods that are presented to the patient's nose. It consists of 3 parts different, with 3 sets of corresponding sticks: an olfactory threshold test, an olfactory discrimination test and an olfactory identification test.
  The final score, out of 48, is the sum of the olfactory threshold, discrimination and identification scores. Normal test values are defined as greater than the tenth percentile of the general population, so the test result is compared to reference values on a chart to determine whether the patient is normosmic, hyposmic or anosmic.
Other: numerical evaluation scale for olfaction — numerical rating scale from 0 (no smell) to 10 (perfect smell)
  Arms: patients with chronic rhinosinusitis with nasal polyps
Other: numerical evaluation scale for nasal obstruction — numerical rating scale from 0 (no freedom of the nasal passages) to 10 (maximum nasal freedom)
  Arms: patients with chronic rhinosinusitis with nasal polyps
Other: nasal outcome test — list of symptoms and social/emotional consequences of rhino-sinusitis. 16 questions that the patient must code from "no problem" to "serious problem" over the last 15 days
Biological: dosage of 17 cytokines — dosage of 17 cytokines : G-CSF, GM-CSF, IFN-γ, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p70), IL-13, IL-17A, MCP-1 (MCAF), MIP-1β,TNF-α

SUMMARY:
Impaired olfaction is one of the major complaints of patients with nasosinus polyposis, with nasal obstruction. In case of failure of medical treatment for patients with polyposis nasosinusal, they may use endoscopic surgery nasosinusal. Before surgery, 73% are hyposmic or anosmic, compared to 43% after surgery. Persistence of hyposmia or anosmia despite the removal of polyps can be explained by mechanisms inflammatory in the mucous membrane of the olfactory cleft. In addition, studies in mice have shown a degeneration of primary olfactory neurons at the level of the olfactory mucosa in connection with directly with TNF alpha, a pro-inflammatory molecule.

ELIGIBILITY:
Inclusion Criteria for patients :

* Patients with nasosinus polyposis requiring nasosinus surgery
* Patient affiliated or entitled to a social security
* signed consent

Inclusion Criteria for control group :

* Patients with an indication for septoplasty
* Patient affiliated or entitled to a social security
* signed consent

Exclusion Criteria for patients :

* Patients with nasosinus polyposis secondary to another disease
* Patients with hyposmia or anosmia prior to naso-sinus polyposis
* Patients with diagnosed neurodegenerative disease
* Patients who are mentally or physically unable to perform olfactory tests
* Patients on anti-TNF-alpha therapy, long-term oral corticosteroid therapy, or other immunomodulatory therapy.

Exclusion Criteria for control group :

* Patients with nasosinus polyposis
* Patients with chronic rhino-sinusitis
* Patients with hyposmia or anosmia
* Patients with diagnosed neurodegenerative disease
* Patients who are mentally or physically unable to perform olfactory tests
* Patients on anti-TNF-alpha therapy, long-term oral corticosteroid therapy, or other immunomodulatory therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
expression rate of TNF-alpha in biopsies | 2 months
  The main evaluation criterion is based on two variables: the expression rate of TNF-alpha in olfactory slit biopsies and the Sniffin Stick test score.
Sniffin Stick test score | 2 months
  The main evaluation criterion is based on two variables: the expression rate of TNF-alpha in olfactory slit biopsies and the Sniffin Stick test score.
  Sniffin Stick test score :
  The final score, out of 48, is the sum of the olfactory threshold (out of 16), discrimination (out of 16) and identification (out of 16) scores.
  Normal test values are defined as greater than the tenth percentile of the general population, so the test result is compared to reference values on a chart to determine whether the patient is normosmic, hyposmic or anosmic.

SECONDARY OUTCOMES:
Olfactory Cleft Endoscopic Score | 2 months
  measured at control and patients. 5 endoscopic feature to be completed :
  * discharge : 0= none or scant clear/thin drainage (normal) ; 1= more abundant, thicker clear/white drainage (not normal but not purulent) ; 2= thicker, more abundant, discolored/purulent drainage.
  * polyps : 0= none ; 1= discrete polyps partially narrowing/blocking the olfactory cleft (<50%) ; 2= discrete polyps completely narrowing/blocking the olfactory cleft (>50%).
  * edema : 0= none ; 1= swelling partially narrowing/blocking the olfactory cleft (<50%) ; 2= swelling completely narrowing/blocking the olfactory cleft (>50%).
  * crusting : 0= none ; 1= mild ; 2= severe
  * scarring : 0= none ; 1= mild ; 2= severe
expression rate of TNF-alpha in polyps | 2 months
  measured at control and patients.
dosage of cytokines G-CSF | 2 months
  measured at control and patients.
dosage of cytokines GM-CSF | 2 months
  measured at control and patients.
dosage of cytokines IFN-γ | 2 months
  measured at control and patients.
dosage of cytokines IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12, IL-13, IL-17A | 2 months
  measured at control and patients.
dosage of cytokines MCP-1 | 2 months
  measured at control and patients.
dosage of cytokines MIP-1β | 2 months
  measured at control and patients.
dosage of cytokines MCAF | 2 months
  measured at control and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marie GAVID, MD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No